CLINICAL TRIAL: NCT00981656
Title: A Phase II Protocol for Patients With Stage T1 Bladder Cancer to Evaluate Selective Bladder Preserving Treatment by Radiation Therapy Concurrent With Radiosensitizing Chemotherapy Following a Thorough Transurethral Surgical Re-Staging
Brief Title: Radiation Therapy and Chemotherapy in Treating Patients With Stage I Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0926; CDR0000654727; NCI-2011-01974 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
Keywords: stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Fluorouracil; Mitomycin; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3DCRT + CT (Experimental): Concurrent three-dimensional conformal radiation therapy (3DCRT) and radiosensitizing chemotherapy (CT) consisting of either cisplatin alone or the combination of mitomycin and 5-fluorouracil. Protocol treatment must begin with 15 weeks after a transurethral resection of the tumor (TURBT).
  Interventions: Drug: cisplatin; Drug: 5-fluorouracil; Drug: Mitomycin; Radiation: Three-Dimensional Conformal Radiation Therapy

INTERVENTIONS:
Drug: cisplatin — 60-minute intravenous (IV) infusion of 15 mg/m^2 on days 1, 2, 3, 15, 16, 17, 29, 30, and 31 of radiation treatment.
Drug: 5-fluorouracil — Continuous IV infusion of 500 mg/m^2/24 hrs for 5 consecutive days during weeks 1 and 4 of radiation treatment.
  Other Names: 5FU
Drug: Mitomycin — IV bolus dose of 12 mg/m^2 on day 1 of radiation treatment.
Radiation: Three-Dimensional Conformal Radiation Therapy — Total dose to the gross bladder volume of 61.2 Gy as 34 daily fractions 5 days/week, for approximately 7 weeks.
  Other Names: 3DCRT; 3D CRT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin, mitomycin C, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with cisplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well radiation therapy given together with chemotherapy works in treating patients with stage I bladder cancer.

DETAILED DESCRIPTION:
After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and annually thereafter until termination of the study.

ELIGIBILITY:
Inclusion criteria

1. Pathologically proven diagnosis of carcinoma of the bladder within 105 days prior to registration.

   • Operable patients whose initial tumor is a primary high grade urothelial carcinoma of the bladder exhibiting histologic evidence of invasion into the lamina propria (disease clinical stage T1) or a high grade stage Ta urothelial carcinoma without hydronephrosis; patients who have involvement of the prostatic urethra with urothelial carcinoma and have no evidence of stromal invasion of the prostate remain eligible. If the patient's initial tumor was a high grade stage Ta urothelial carcinoma then his/her recurrent tumor must be a high grade stage T1 urothelial carcinoma to be eligible.
2. Patients must have a high grade urothelial carcinoma stage Ta or T1 that has recurred within 540 days after completion of the initial treatment [TURBT and intravesical Bacillus Calmette Guerin (BCG) immunotherapy] or on initial presentation with a T1 high grade tumor, the participating urologist judged BCG therapy is contraindicated or unsuitable because the patient is found to be intolerant of BCG therapy or because this patient may be immuno-compromised in ways other than that mentioned in Exclusion Criteria 2.8 or because the patient refuses BCG therapy.
3. With the presentations as described in Section 2, the participating urologist judges that the standard next therapy, based on present urologic guidelines for this patient, is radical cystectomy.
4. If radiologic evaluation of a lymph node is interpreted as "positive", this must be evaluated further either by lymphadenectomy or by percutaneous needle biopsy. Patients with histologically or cytologically confirmed node metastases will not be eligible.
5. Patients must have an adequately functioning bladder as judged by the participating urologist and radiation oncologist and have undergone a re-staging TURBT by the participating urologist that showed (or was present in the outside pathology specimen) a high grade stage Ta or T1 tumor with uninvolved muscularis propria in the specimen and, if on prostatic urethral biopsy mucosal carcinoma is present, there is no evidence on biopsy in the prostatic stroma of tumor invasion.
6. Patient must be considered able to tolerate systemic chemotherapy combined with pelvic radiation therapy, and a radical cystectomy (if necessary) by the joint agreement of the participating urologist, radiation oncologist, and medical oncologist.
7. Appropriate stage for protocol entry, based upon the following minimum diagnostic workup within 60 days prior to registration:

   • History/physical examination including weight, performance data, body surface area
8. Zubrod Performance Status ≤ 1
9. Age ≥ 18
10. Complete blood count (CBC)/differential obtained no more than 30 days prior to registration on study, with adequate bone marrow function defined as follows:

    * White blood cell count (WBC) ≥ 4,000/ml
    * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
    * Platelets ≥ 100,000 cells/mm3
    * Hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable.)
11. If the patient is to be treated with cisplatin, the serum creatinine should be ≤ 1.5 mg%; serum bilirubin of ≤ 2.0 mg%
12. Glomerular filtration rate (GFR) > 25 ml/min [For patients receiving cisplatin, GFR ≥ 60 ml/min]
13. Serum pregnancy test for female patients of childbearing potential, ≤ 72 hours prior to study entry; women of childbearing potential and male participants must practice adequate contraception.
14. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria

1. Evidence of tumor-related hydronephrosis
2. Evidence of distant metastases or histologically or cytologically proven lymph node metastases
3. Prior systemic chemotherapy for bladder cancer; prior chemotherapy for a different cancer is allowable
4. A prior or concurrent malignancy of any other site or histology unless the patient has been disease-free for ≥ 5 years except for non-melanoma skin cancer and/or stage T1a prostate cancer or carcinoma in situ of the uterine cervix or a urothelial carcinoma of the upper urinary tract stage pTa, pTis or pT1 that has not been free of disease after treatment for more than a 2-year period
5. Patients with pN+ or > T1 disease or who have not had a visibly complete TURBT
6. Patients receiving any drugs that have potential nephrotoxicity or ototoxicity (such as an aminoglycoside)
7. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * Transmural myocardial infarction within the last 6 months;
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * Acquired Immune Deficiency Syndrome (AIDS) based upon the current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
9. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
10. Prior allergic reaction to the study drugs (cisplatin, mitomycin, 5FU) involved in this

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William U. Shipley, MD, FACR, Principal Investigator — Massachusetts General Hospital
Locations (13):
- United States (13):
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont

REFERENCES:
- [Derived] Dahl DM, Rodgers JP, Shipley WU, Michaelson MD, Wu CL, Parker W, Jani AB, Cury FL, Hudes RS, Michalski JM, Hartford AC, Song D, Citrin DE, Karrison TG, Sandler HM, Feng FY, Efstathiou JA. Bladder-Preserving Trimodality Treatment for High-Grade T1 Bladder Cancer: Results From Phase II Protocol NRG Oncology/RTOG 0926. J Clin Oncol. 2024 Dec;42(34):4095-4102. doi: 10.1200/JCO.23.02510. Epub 2024 Sep 3. PMID 39226514

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3DCRT + CT
Started | 37
Eligible and Started Study Treatment | 34
Completed (Participants contributing data to results are considered to have completed the study.) | 34
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Did not start protocol treatment | 2

BASELINE CHARACTERISTICS:
Population: Eligible participants who started study treatment
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  Years: ≤ 59 | 4
  Years: 60-69 | 12
  Years: 70-79 | 14
  Years: ≥ 80 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Zubrod [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 29
    1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From Radical Cystectomy at 3 Years
Description: The number of participants who did not undergo a radical cystectomy within three years divided by the number of analyzed participants, presented with the 97.5% lower bound.
Time Frame: Three years from registration
Population: Eligible participants who started study treatment
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 88.2 [72.5 to NA] — An upper bound was not calculated per protocol. (All alpha is used for the lower bound.)
Statistical Analysis 1: Comparison: 3DCRT + CT; Null hypothesis = this treatment will result in 75% of participants free from radical cystectomy at 3 years. A lower confidence bound of 60% will be promising enough to pursue this regimen further. A sample size of 33 analyzable patients provides a one-sided 97.5% lower bound of 60% relative to the hypothesized 75%. In terms of type I error, this design provides a 2.5% chance of observing a 3-year percentage less than 60% if the true rate is 75%; Test type: Other — No testing is done, conclusions are made based on the confidence interval; If the lower confidence interval (CI) limit was above 60% then the regimen would be considered promising enough to warrant further study for this treatment regimen. If the lower limit was below 25% then the treatment would not be considered worthy of further study. If the lower limit fell between 25% and 60%, the investigators would consider the possibility of further investigation

2. Secondary Outcome: Percentage of Participants Free From Radical Cystectomy at 5 Years
Description: The number of participants who did not undergo a radical cystectomy within five years divided by the number of analyzed participants.
Time Frame: Five years from registration
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 88.2 [72.5 to 96.7]

3. Secondary Outcome: Percent of Participants With Distant Disease Progression at 3 Years
Description: Distant disease progression is defined as the first appearance of disease in a non-regional lymph node, solid organ or bone. Time to distant disease progression is defined as time from registration to the date of first distant disease progression, last known follow-up (censored), or death without distant disease progression (competing risk). Distant disease progression rate is estimated using the cumulative incidence method.
Time Frame: From registration to three years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 12.3 [3.8 to 26.3]

4. Secondary Outcome: Percent of Participants With Distant Disease Progression at 5 Years
Description: as for outcome 3
Time Frame: From registration to five years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 18.7 [7.4 to 34.0]

5. Secondary Outcome: Percentage of Participants With Progression to Tumor Stage T2 or Greater at 3 Years
Description: Primary tumor stage T2 = tumor invades muscle; T3 = tumor invades perivesical tissue; T4 = tumor invades any of the following: prostate, uterus, vagina, pelvic wall, abdominal wall. Time to progression is defined as time from registration to the date of first progression, last known follow-up (censored), or death without tumor progression (competing risk). Tumor progression rates was to be estimated using the cumulative incidence method.
Time Frame: From registration to three years
Population: T-stage was not collected on follow-up forms and therefore this outcome measure could not be not analyzed.
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Progression to Tumor Stage T2 or Greater at 5 Years
Description: Primary tumor stage T2 = tumor invades muscle; T3 = tumor invades perivesical tissue; T4 = tumor invades any of the following: prostate, uterus, vagina, pelvic wall, abdominal wall. Time to progression is defined as time from registration to the date of first progression, last known follow-up (censored), or death without tumor progression (competing risk). Tumor progression rate was to be estimated using the cumulative incidence method.
Time Frame: From registration to five years
Population: T-stage was not collected on follow-up forms and therefore this outcome measure cab not be not analyzed.
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants Who Have Died From Bladder Cancer at 5 Years (Disease-specific Survival)
Description: Time to death from bladder cancer is defined as time from registration to death from bladder cancer, last known follow-up (censored), or death from other cause (competing risk). More specifically, death absent a distant metastasis, death from non-bladder cancer, and death absent local recurrence comprise the competing risk. Death from bladder cancer rate is estimated using the cumulative incidence method.
Time Frame: From registration to five years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 25.1 [11.5 to 41.3]

8. Secondary Outcome: Percentage of Participants Alive at 3 Years
Description: Overall survival time is defined as time from registration to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: From registration to three years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 69.2 [53.3 to 85.2]

9. Secondary Outcome: Percentage of Participants Alive at 5 Years
Description: as for outcome 8
Time Frame: From registration to five years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 56.4 [39.1 to 73.7]

10. Secondary Outcome: Distribution of Participants by Highest Grade Adverse Event
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 4 grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: Adverse events are evaluated 8-10 weeks after end of study treatment (approximately 7 weeks), then every 3 months for one year, every 4 months for one year, every 6 months for 3 years, then annually. Maximum follow-up at time of reporting was 8.6 years.
Population: Eligible participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
Participants
  Grade 1 | 2
  Grade 2 | 9
  Grade 3 | 20
  Grade 4 | 2
  Grade 5 | 0

11. Secondary Outcome: Percentage of Participants With Local Recurrence at 3 Years
Description: Time to local recurrence is defined as time from registration to the date of first local recurrence, last known follow-up (censored), or death without local recurrence (competing risk). Local recurrence rate is estimated using the cumulative incidence method.
Time Frame: From registration to three years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 34
percentage of participants | 32.5 [17.4 to 48.6]

12. Secondary Outcome: American Urological Association Total Symptom Score at Baseline and at 3 Years
Description: The American Urological Association Total symptom score measures the severity of enlarged prostate symptoms. Possible scores range from 0 to 35, with higher scores indicating worse symptoms.
Time Frame: Baseline and 3 years
Population: Eligible participants who started study treatment and have baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3DCRT + CT
Number analyzed (Participants) | 32
units on a scale
  Baseline | 9.84 (6.47)
  Three years: number analyzed (Participants) | 9
  Three years | 12.00 (9.25)

ADVERSE EVENTS:
Time Frame: Adverse events are evaluated 8-10 weeks after completion of study treatment (approximately 7 weeks), then every 3 months for one year, every 4 months for one year, every 6 months for three years, then annually. Maximum follow-up at time of reporting was 8.6 years.
Arm/Group | 3DCRT + CT
All-Cause Mortality (participants affected / at risk) | 15/34
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3DCRT + CT (N=34)
Atrial fibrillation (Cardiac disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3DCRT + CT (N=34)
Anemia (Blood and lymphatic system disorders) | 20
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 21
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6
Hemorrhoids (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Rectal hemorrhage (Gastrointestinal disorders) | 2
Chills (General disorders) | 4
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 28
Fever (General disorders) | 4
Pain (General disorders) | 6
Bladder infection (Infections and infestations) | 2
Mucosal infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 12
INR increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 14
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Bladder spasm (Renal and urinary disorders) | 5
Cystitis noninfective (Renal and urinary disorders) | 8
Hematuria (Renal and urinary disorders) | 11
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 12
Urinary frequency (Renal and urinary disorders) | 24
Urinary incontinence (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 5
Urinary urgency (Renal and urinary disorders) | 11
Erectile dysfunction (Reproductive system and breast disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT00981656/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT00981656/ICF_001.pdf